CLINICAL TRIAL: NCT02954484
Title: Outcomes Of Perioperative Pregabalin On Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Outcomes Of Perioperative Pregabalin On Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190514
Record Dates: First submitted 2016-10-20; First posted 2016-11-03 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2016-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Etoricoxib; Acetaminophen; Morphine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREGABALIN (Active Comparator): All subjects receive intravenous PCA morphine, paracetamol 1g po six hourly and etoricoxib 120mg po once daily. Subjects receive pregabalin 75mg orally preoperatively followed by 75mg at night for two days. During surgery, patients received general anaesthesia with femoral nerve block on the side of surgery.
  Interventions: Drug: pregabalin; Drug: Etoricoxib; Drug: paracetamol; Drug: Morphine; Drug: Ropivacaine
- PLACEBO (Placebo Comparator): All subjects receive intravenous PCA morphine, paracetamol 1g po six hourly and etoricoxib 120mg po once daily. Subjects receive either placebo tablet (of identical appearance to pregabalin) orally preoperatively followed by 75mg at night for two days. During surgery, patients received general anaesthesia with femoral nerve block on the side of surgery.
  Interventions: Drug: Placebo; Drug: Etoricoxib; Drug: paracetamol; Drug: Morphine; Drug: Ropivacaine

INTERVENTIONS:
Drug: pregabalin — see arm/group description. Lyrica manufacture site: Pfizer Manufacturing Deutschland GmbH, Freiburg, Germany.
  Other Names: Lyrica (Pfizer Pte Ltd, Singapore)
  Arms: PREGABALIN
Drug: Placebo — Placebo capsule containing lactose and MCC (no active ingredients).
  Other Names: Manufactured by Beacons Pharmaceuticals Pte Ltd, Singapore.
  Arms: PLACEBO
Drug: Etoricoxib — Etoricoxib 120mg per oral once daily on postoperative days 1,2,3. 'Arcoxia' manufacture site: MSD International GMBH, Singapore
  Other Names: 'Arcoxia'
Drug: paracetamol — Paracetamol 1g per oral 6hourly on postoperative days 1,2,3. Manufacture site: SM Pharmaceuticals, Malaysia
  Other Names: acetaminophen
Drug: Morphine — patient-controlled analgesia intravenous morphine sulphate on postoperative days 1,2,3.
  Manufacture site: Hameln Pharma Plus GMBH, Hameln, Germany
Drug: Ropivacaine — Femoral block with ropivacaine 0.5% 30mls. Ropivacaine manufacture site: AstraZeneva AB, Sweden
  Other Names: 'Naropin'

SUMMARY:
This study aims to provide high quality evidence from a double-blinded, randomized controlled trial on the efficacy of perioperative pregabalin in reducing morphine requirements, improving pain scores and reducing chronic neuropathic pain when compared with placebo for primary total knee arthroplasty. It hence aims to improve on choice of analgesia adjuncts for total knee arthroplasty.

DETAILED DESCRIPTION:
Aims:

Whether pregabalin given preoperatively and for one week postoperatively in addition to patient-controlled analgesia (PCA) morphine is effective in reducing morphine requirements, improving pain scores and reducing chronic neuropathic pain when compared with placebo for primary total knee arthroplasty.

Methodology:

A single-centre double-blind randomized controlled trial in patients undergoing primary total knee arthroplasty. All subjects receive PCA morphine, paracetamol 1g every six hours, etoricoxib 120mg once daily postoperatively. Subjects receive either pregabalin 75mg po preoperatively followed by 75mg OM and 25mg ON for two days postoperatively or matching placebo. The primary outcome is cumulative morphine consumption at 72 hr following surgery. Secondary outcome measures included pain scores, knee range of motion and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary total knee arthroplasty

Exclusion Criteria:

* revision or bilateral arthroplasty, significant renal or hepatic impairment, documented allergy or intolerance to NSAIDs, paracetamol, morphine or pregabalin, chronic pain syndrome treated with chronic opioids, obstructive sleep apnea not treated with continuous positive airway pressure, seizures, breastfeeding, inability to use patient-controlled analgesia.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption at 72 hours postoperatively | 72 hours postoperatively

SECONDARY OUTCOMES:
Functional scores: SF-36v2 at 3 months and 6 months postoperatively | 3 months and 6 months postoperatively
Functional scores: Knee Society Score at 3 months and 6 months postoperatively | 3 months and 6 months postoperatively
Functional scores: WOMAC at 3 months and 6 months postoperatively | 3 months and 6 months postoperatively
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Knee range of motion at 3 months and 6 months postoperatively | 3 months and 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: lingaraj krishna, frcs (Orth), Principal Investigator — National University Health System, Singapore

IPD SHARING:
Plan to Share IPD: No